CLINICAL TRIAL: NCT00501215
Title: Pilot Study on the Effect of Parathyroidectomy on Sleep
Brief Title: Effect of Parathyroidectomy on Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0220; NCI-2010-00658 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Hyperparathyroidism
Keywords: Primary Hyperparathyroidism; PHPT; Parathyroidectomy; Polysomnogram; PSG; Sleep Quality; Interview
MeSH Terms: conditions — Hyperparathyroidism; Hyperparathyroidism, Primary; Sleep Initiation and Maintenance Disorders | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parathyroidectomy + Observation (Experimental)
  Interventions: Procedure: Parathyroid Surgery; Behavioral: Telephone Interview; Behavioral: Polysomnography (PSG)
- Observation Alone (Other)
  Interventions: Behavioral: Telephone Interview; Procedure: Parathyroid Surgery; Behavioral: Polysomnography (PSG)

INTERVENTIONS:
Procedure: Parathyroid Surgery — Parathyroid surgery 1-3 weeks after the first PSG.
  Arms: Parathyroidectomy + Observation
Behavioral: Telephone Interview — Interview about sleep quality lasting 15-20 minutes.
Procedure: Parathyroid Surgery — Parathyroid surgery after completing the second PSG and after the study participation ends.
  Arms: Observation Alone
Behavioral: Polysomnography (PSG) — 2 overnight sleep tests
  Group 1: First PSG 1-3 weeks before surgery + Second PSG 6-8 weeks after surgery
  Group 2: First PSG 1-3 weeks before phone interview + Second PSG 6-8 weeks after phone interview
  Other Names: nocturnal polysomnography; sleep study; sleep test; sleep survey; sleep evaluation

SUMMARY:
Primary hyperparathyroidism (PHPT) is an endocrine disorder that disrupts calcium metabolism and has a broad range of clinical manifestations. With respect to the nonclassic, subjective symptoms that have been reported to be associated with PHPT, such as sleep disturbance, neurocognitive dysfunction, mood disturbance, fatigue, and decreased quality of life, there is a lack of objective data on the extent to which these symptoms are affected by parathyroidectomy.

There have been reports of improvements in sleep in patients following parathyroidectomy, but these have been based solely on subjective sleep surveys. To date, there are no published studies on objective sleep evaluations of patients with PHPT. The overall goals of this protocol are to ascertain the feasibility of performing sleep studies on patients with PHPT, and to obtain pilot data on the effects of parathyroidectomy on those sleep studies.

It is hypothesized that it will be feasible to evaluate sleep parameters in patients with PHPT in the M. D. Anderson Sleep Center. Towards testing this hypothesis, the specific aims are:

Specific Aim 1: To assess the feasibility of using nocturnal polysomnography (PSG) to evaluate the primary outcome measure of total sleep time.

Specific Aim 2: To assess the feasibility of using nocturnal polysomnography (PSG) to evaluate the secondary outcome measures of sleep architecture, arousal index, sleep efficiency, wake after sleep onset, and sleep onset latency in patients with PHPT.

Specific Aim 3: To assess the feasibility of evaluating the secondary outcome measures of subjective sleepiness as tested with the Epworth Sleepiness Scale (ESS), and of sleep quality as tested with the Brief Sleep Disturbance Scale (BSDS) in patients with PHPT.

Specific Aim 4: To assess the feasibility using a randomized "wait-list"-control design to assess the effects of parathyroidectomy on sleep measures obtained with nocturnal PSG.

DETAILED DESCRIPTION:
Screening Test:

To be eligible to take part in this study, women who are able to have children must have a negative blood (about 1 teaspoon) pregnancy test.

Study Groups:

If you are found to be eligible to take part in this study and you agree to take part, you will be randomly assigned (as in the toss of a coin) to 1 of 2 groups. There is an equal chance that you will be assigned to either group. One group (the 'Surgical' Group) will receive the parathyroid surgery and "observation" (the review of blood tests by the study doctor) during the course of the study. The other group (the 'Observation' Group) will receive observation alone, and then surgery after their study participation ends.

All participants will have 2 overnight sleep tests (called "polysomnograms" -- PSGs) and a telephone interview on sleep quality.

The Surgical Group will have their first PSG, and then 1-3 weeks later their surgery and a telephone interview will be performed. (For the surgery, a separate informed consent form will be signed that will describe the procedure in detail.) About 6-8 weeks after surgery, a second PSG will be performed.

The Observation Group will have their first PSG, and then a telephone interview 1-3 weeks later. At 6-8 weeks after the interview, a second PSG will be performed. The Observation Group participants will be offered to have their parathyroid surgery soon after they complete their second PSG (after their 7-11 week participation in this study is over).

Sleep Quality Interview:

For the telephone interview, a research staff member will call you at home to ask you to discuss 6 questions about the quality of your sleep. It should take about 15-20 minutes.

Polysomnography:

A PSG is a standard test for evaluating sleep. However, patients with PHPT do not routinely receive PSGs as part of their standard care.

PSGs use many measurements made while the participant is asleep. Sensors on the body record information about a person's sleep stages, body position, blood oxygen levels, breathing, muscle tone, heart rate, snoring, and general sleep behavior.

Electroencephalogram (EEG) sensors will be placed on your scalp and face in order to measure what 'stage' of sleep you are in. Electrocardiogram (ECG) sensors will be placed on your chest to monitor your heartbeat. A small probe will rest just inside your nostrils in order to measure your breathing and airflow. A snoring sensor will be taped on your neck. Elastic straps will be placed around your chest and abdomen (midsection), which will measure your breathing effort. Sensors will be placed on both of your shins in order to measure your leg movements. A sensor will be taped onto your fingertip in order to measure your blood oxygen levels.

Audio and video recordings will be made of your sleep in order to monitor your body positions and to record any sleep disturbances and/or restless movements that may occur.

For both of the PSGs, you will arrive at the M. D. Anderson Sleep Center at about 7:30 p.m. You will complete a questionnaire about your sleep the night before and your activities during that day. You will also complete a questionnaire that asks about any 'dozing off' habits you may have. It should take about 10-15 minutes to complete the 2 questionnaires. You will be taken to a sleep room, which will be quiet and darkened. A registered PSG technologist will place the sensors on your body. You will be allowed to sleep until your usual wake-up time, as noted on your sleep diary. Soon after you wake up, the sensors will be removed. You will complete a third questionnaire about your night's sleep. This last questionnaire should take about 5-10 minutes to complete. You will be able to leave shortly after completing the questionnaire.

If you normal sleep during the day, the study staff will arrange the sleep study to happen around your usual sleeping and waking times.

Sleep Diaries:

For the 7 days before each PSG, you will complete a sleep diary. In the diary, you will record information about the quality and amount of your sleep. You will bring the sleep diary to the Sleep Center on the days of your PSGs.

Biomarker Testing:

Blood (about 4 teaspoons each time) will be drawn earlier in the day of your PSG, before you have the PSG performed. This blood will be used to measure certain biomarkers that will be compared with the results of your PSGs and questionnaires. These biomarkers include the levels of calcium, parathyroid hormone (PTH), and vitamin D in your blood.

Possible Crossover to Surgical Group:

If you are in the Observation Group and your blood tests show very high calcium levels, you will be offered parathyroid surgery as soon as reasonably possible.

Also, if you are in the Observation Group and you start experiencing worsening symptoms that may mean kidney stones (such as abdominal pain and/or blood in the urine) or inflammation of the pancreas (such as abdominal pain, nausea, vomiting, fever, and/or chills), your condition will be evaluated and treated. You will then be offered parathyroid surgery as soon as reasonably possible. At 6-8 weeks after your parathyroid surgery, you will have your second PSG.

Sleep Test Results:

You will be able to receive a copy of your PSG results. If the results show any sleep disorders and/or other medical disorders, you will referred for standard treatment.

The results of the PSG will not affect your PHPT treatment in any way.

Length of Study:

After your second PSG, your participation in this study will be over.

This is an investigational study. Using PSGs for this purpose in patients with PHPT is considered experimental.

Up to 12 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Be diagnosed with PHPT (inappropriate PTH level in the setting of a high or high-normal serum calcium level greater than or equal to 10.0 mg/dL).
2. Have at least one of the following symptoms affecting sleep: a) not feeling refreshed on awakening b) difficulty falling asleep c) waking up during the night d) have difficulty falling back asleep at night after awakening e) waking up too early in the morning f) excessive sleepiness during the day
3. Be considered an appropriate surgical candidate.
4. Be older than 21 years of age.
5. Female participants of childbearing potential must have a negative pregnancy test (urinary or serum beta-HCG).

Exclusion Criteria:

1. Have a known major sleep disorder documented by prior diagnosis, such as: a) sleep disordered breathing b) narcolepsy c) periodic limb movement disorder d) parasomnias
2. Have any other functional tumors if they have familial Multiple Endocrine Neoplasia Syndrome 1 or 2 (MEN 1 or MEN 2).
3. Patients with a calcium level greater than 13mg/dL.
4. Patients with recent history of kidney stones.
5. Patients with recent history of pancreatitis

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-05-25 (Actual); Primary Completion 2017-07-09 (Actual); Study Completion 2017-07-09 (Actual)

PRIMARY OUTCOMES:
Total sleep time | Before and After Intervention

SECONDARY OUTCOMES:
Overnight sleep test to measure effect of treatment with parathyroidectomy may have on patients' sleep. | First set of tests (baseline) will occur within 1-3 weeks prior to intervention/assessment, and the second set of tests will occur 6-8 weeks after the intervention/assessment.
Effectiveness of 2 sleep-related questionnaires to measure certain sleep-related factors in patients with PHPT. | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Nancy D. Perrier, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Morris GS, Grubbs EG, Hearon CM, Gantela S, Lee JE, Evans DB, Holmes HM, Busaidy NL, Jimenez C, Perrier ND. Parathyroidectomy improves functional capacity in "asymptomatic" older patients with primary hyperparathyroidism: a randomized control trial. Ann Surg. 2010 May;251(5):832-7. doi: 10.1097/SLA.0b013e3181d76bb3. PMID 20395857
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org